CLINICAL TRIAL: NCT02199353
Title: Effectiveness of A Therapy Programme Based On The Reestablishment of Cognitive Functions on The Independence of Patients With Dementia Performing Activities of Daily Living - A Pilot Study
Brief Title: Occupational Therapy Programme of Patients With Dementia Performing Activities of Daily Living
Acronym: OTSALD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, MARIA JIMENEZ PALOMARES, Profesor of Occupational Therapy, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 46/2012
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Dementia
Keywords: Activities of daily living, Occupational Therapy, Dementia
MeSH Terms: conditions — Dementia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation of Activities Daily Living (Experimental): The experimental group received the Stimulation of Activities of Daily Living (SADL) programme which is a new treatment approach created by the authors of this study for the training of activities of daily living (ADL) through cognitive intervention. The programme is based on the reestablishment of the cognitive functions implied in the performance of basic activities of daily living.
  The sequence of the sessions was always the same, varying the activities, subject, cognitive functions and BADL to work on. Each session started with an activity of temporal and space orientation, continued with the performance of the specific activity of the session and finished with a reminiscence activity.
  The treatment was applied twice a week (Tuesday and Thursday) for 45 minutes during 5 weeks.
  Interventions: Other: Stimulation of Activities Daily Living
- Conventional ADLoccupational therapy (Active Comparator): The control group treatment was based on a conventional occupational therapy intervention for the management of ADL deficits. The compensation approach was used and environment modifications and simplification of activities were applied as the intervention method.
  The treatment was carried out twice a week (Tuesday and Thursday) for 45 minutes during 5 weeks.
  Interventions: Other: Conventional ADLOccupational Therapy

INTERVENTIONS:
Other: Stimulation of Activities Daily Living — Experimental group: SADL programme which is a new treatment approach created by the authors of this study for the training of ADL through cognitive intervention. The programme is based on the reestablishment of the cognitive functions implied in the performance of basic activities of daily living.
  The treatment was carried out twice a week (Tuesday and Thursday) for 45 minutes during 5 weeks.
  Other Names: Occupational therapy
  Arms: Stimulation of Activities Daily Living
Other: Conventional ADLOccupational Therapy — Control group treatment: conventional occupational therapy intervention for the management of ADL deficits. The compensation approach was used and environment modifications and simplification of activities were applied as the intervention method.
  The treatment was carried out twice a week (Tuesday and Thursday) for 45 minutes during 5 weeks.
  Arms: Conventional ADLoccupational therapy

SUMMARY:
To assess the effectiveness of the Stimulation of Activities of Daily Living (SADL) Occupational Therapy programme on the independence of ADL by persons with dementia who are institutionalized. This programme is based on the recovery of the cognitive functions.

DETAILED DESCRIPTION:
This study is a longitudinal and prospective clinical trial approved by the bioethics Commission of the University of Extremadura. 58 senior citizens institutionalized with dementia in residential homes in Extremadura (Spain) received a treatment focusing on activities of daily living with the SADL programme and with conventional occupational therapy during 5 weeks. The studied variables were the cognitive level and the independence level performing ADL. The variables were measured by an occupational therapist independent to the study at baseline, after 5 weeks of experimental treatment and 6 weeks after the treatment was completed. The standardized tests used were Barthel Index, Lobo's Cognoscitive mini test, Lawton and Brody Scale and Global Deterioration Scale (GDS).

ELIGIBILITY:
Inclusion Criteria:

* Institutionalization in residential homes at least 6 months before the commencement of the study.
* Diagnosis of dementia for at least one year according to the Diagnostic and Statistical Manual of Mental Disorders (DMS IV) criteria.
* Over 60 years old.
* Barthel Index scores greater than or equal to 40%.
* Lobo´s Cognitive Mini Test scores greater than or equal to 15 points.
* To be included in the BADL intervention programme of Occupational therapy in the previous 6 months and to have the informed consent signed by the legal tutor.

Exclusion Criteria:

* To present psychological or behavior symptoms diagnosed by a doctor.
* Barthel Index scores less than 40%
* Not being included in the BADL intervention programme of Occupational therapy in the previous 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Dependency level | after 5 weeks of treatment and after 6 weeks of follow up
  In order to assess the basic activities of daily living (BADL), Barthel Index published in 1.965 by Mahoney y Barthel was applied. This scale provides information at a global level with the general scores (dependence level) and at a specific level with each item's score. A score of less than 20 means total dependence, 20-35 scores mean severe dependence, 40-55 scores mean moderate dependence, equal or over 60 means mild dependency and 100 means independence. This allows the assessment of any changes in each basic activity area evaluated with this scale

SECONDARY OUTCOMES:
Cognitive level. | After 5 weeks of treatment and after 6 weeks of follow up
  To assess the cognitive level and guarantee the homogeneity of the sample, the adapted and validated Spanish version of the Mini Mental Status Examination (MMSE) test by Lobo et al was used. The Global Deterioration Scale (GDS) designed by Reisberg et al was also used to determine the deterioration level.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jimenez, Professor, Principal Investigator — University of Extremadura
Locations (1):
- 'CARE' elderly residential homes, Cáceres, Cáceres, Spain